CLINICAL TRIAL: NCT00610753
Title: Family Therapy in the Treatment of Adolescent Anorexia Nervosa
Brief Title: Comparison of Two Types of Family Therapy in the Treatment of Adolescent Anorexia Nervosa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, William Stewart Agras, Professor Emeritus, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SU-12132007-933; 5 U01 MH076290; SPO#33857; 5U01MH076290 (NIH)
Record Dates: First submitted 2008-01-25; First posted 2008-02-08 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia nervosa; Adolescents; Family therapy
MeSH Terms: conditions — Anorexia Nervosa | interventions — Family Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Family Behavioral Therapy (Experimental): This intervention focuses on counseling the parents (and other family members) on refeeding their child. When weight is being steadily regained the focus of therapy shifts to allow the child more independence.
  Interventions: Behavioral: Family Behavior Therapy
- Systems Family Therapy (Active Comparator): This therapy focuses primarily on clarifying psychological processes within the family.
  Interventions: Behavioral: Systems Family Therapy

INTERVENTIONS:
Behavioral: Family Behavior Therapy — This treatment is usually delivered in two phases: In the first phase there is an initial investigation of family behavior around feeding using a family meal followed by family therapy focused on enhancing feeding of the anorexic child in order to promote weight gain. In the second phase, once weight gain is well established the adolescent is given greater autonomy over feeding and in later sessions over other issues.
  Other Names: Maudsley Family Therapy
  Arms: Family Behavioral Therapy
Behavioral: Systems Family Therapy — This therapy is applied in three phases. 1. In the first 2 or 3-sessions the treatment is explained to the family and an initial examination of family issues begins. 2. In the second phase family interactions and psychological processes are explored with clarification for family members. 3. In the third phase knowledge of family patterns is refined aiming for behavior change.
  Other Names: Family Therapy
  Arms: Systems Family Therapy

SUMMARY:
This study will compare the effectiveness of two different family treatments for the treatment of adolescent anorexia nervosa.

DETAILED DESCRIPTION:
The long-term objective of this study is to enhance the treatment and outcome of anorexia nervosa (AN). Research on the treatment of AN has lagged that of other conditions, even other eating disorders such as bulimia nervosa. The focus of this study is on adolescent AN. Successful early treatment is likely to reduce the prevalence of chronic AN with its high rates of morbidity and mortality and high health care costs. The most promising treatment for adolescent AN is a specific form of family therapy called behavioral family therapy (BFT). This treatment is focused on the disordered eating behavior that characterizes AN and enables parents to refeed their child. Although there have been several small scale studies of BFT there has been no controlled comparison with another form of family therapy. Therefore we propose to use systems family therapy (SFT) which has been developed to represent the type of family therapy practiced in the community.

One hundred and sixty adolescents of both genders aged 12-18 years meeting DSM-IV criteria for anorexia nervosa will be entered to the study. Recruitment is projected to extend for 2 years. Participants will be randomly allocated to one of the two types of family therapy. Family therapy will be given for 36-weeks. For the purpose of the present study, patients will be followed for 12-months after the end of family treatment. Hence, each family will participate for approximately 2-years, with a total participation time of some 40-hours. In a sub-study blood will be drawn from those volunteering for genetic analysis focusing on the subset of non-responders to treatments.

ELIGIBILITY:
Inclusion Criteria:Diagnosis of anorexia nervosa with Ideal Body Weight >75% Exclusion Criteria:Current psychotic illness or mental retardation that would prohibit the use of psychotherapy Medically unstable for outpatient treatment

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 164 (Actual)
Dates: Start 2006-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Percent Ideal Body Weight (%IBW) | 9-months and 21-months
  Patients weighed in gowns on calibrated balance beam machines and height assessed with a stadiometer. Percent Ideal Body Weight calculated on a study designed calculator.

SECONDARY OUTCOMES:
Eating Disorder Psychopathology | 9 months and 21 months
  Eating Disorders Examination obtained in a standardized interview assessing: Binge eating, purging, weight and shape concerns. Assessed as the global measure.

CONTACTS AND LOCATIONS:
Overall Officials: William Stewart Agras, Principal Investigator — Stanford University
Locations (7):
- United States (6):
  - UCSD Center for Eating Disorder Treatment & Research, San Diego, California
  - Stanford University School of Medicine, Stanford, California
  - Sheppard-Pratt Health System, Baltimore, Maryland
  - Washington University, Department of Psychiatry, St Louis, Missouri
  - Department of Psychiatry, Cornell University, White Plains, New York
  - Laureate Psychiatric Clinic & Hospital, Tulsa, Oklahoma
- Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Lock J, Brandt H, Woodside B, Agras S, Halmi WK, Johnson C, Kaye W, Wilfley D. Challenges in conducting a multi-site randomized clinical trial comparing treatments for adolescent anorexia nervosa. Int J Eat Disord. 2012 Mar;45(2):202-13. doi: 10.1002/eat.20923. Epub 2011 Apr 14. PMID 21495052
- [Derived] Sadeh-Sharvit S, Arnow KD, Osipov L, Lock JD, Jo B, Pajarito S, Brandt H, Dodge E, Halmi KA, Johnson C, Kaye W, Wilfley D, Agras WS. Are parental self-efficacy and family flexibility mediators of treatment for anorexia nervosa? Int J Eat Disord. 2018 Mar;51(3):275-280. doi: 10.1002/eat.22826. Epub 2018 Jan 4. PMID 29314160
- [Derived] Agras WS, Lock J, Brandt H, Bryson SW, Dodge E, Halmi KA, Jo B, Johnson C, Kaye W, Wilfley D, Woodside B. Comparison of 2 family therapies for adolescent anorexia nervosa: a randomized parallel trial. JAMA Psychiatry. 2014 Nov;71(11):1279-86. doi: 10.1001/jamapsychiatry.2014.1025. PMID 25250660